CLINICAL TRIAL: NCT06082310
Title: Biking vs. Running HIIT in Men With Overweight/Obesity: Impact on Oxygen Consumption, Substrate Utilization and Appetite
Brief Title: Biking vs. Running: Comparison of EPOC, Substrate Oxidation, Appetite and Energy Intakes in Men With Overweight/Obesity.
Acronym: BIKERUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Collaborators: CREPS Auvergne-Rhône-Alpes de Vichy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00012476-2022-22-09-199
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Overweight and Obesity
Keywords: Modalities; High-intensity interval exercise; Substrate oxidation; Appetite; Energy Intakes; Enjoyment
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data collected on the volunteers will be made anonymous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training - Biking (HIITBIKE) (Experimental): Cycling exercise: 5 min warm-up + 9-12 x [45 seconds at 80% of HRmax followed by 1 minute 30 seconds of active recovery at a power equivalent to 40% of HRmax].
  Interventions: Other: Exercise
- High Intensity Interval Training - Running (HIITRUN) (Experimental): Running exercise: 5 min warm-up + 9-12 x [45 seconds at 80% of HRmax followed by 1 minute 30 seconds of active recovery at a treadmill speed equivalent to 40% of HRmax].
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Two HIIT modalities

SUMMARY:
The management of obesity involves hygienic and dietary measures that include appropriate nutrition and an increase in physical activity (PA). Among the various PA modalities that can be recommended, High-Intensity Interval Training (HIIT) is now recognized as a fun and effective program for promoting fat loss. A meta-analysis conducted by our team suggests a potential influence of the mode of HIIT practice (cycling vs. running) on fat mass (FM) loss. In order to better understand the metabolic adaptations following this type of practice, the investigators propose to compare two isoenergetic HIIT sessions (cycling vs. running) in overweight or obese subjects. The objective is to compare post-recovery (+2h) oxygen consumption, substrate utilization, concurrent energy expenditure and post 24h energy intakes.

DETAILED DESCRIPTION:
Overweight/obesity, and more specifically intra-abdominal fat mass (FM), are strongly correlated with the development of cardiovascular diseases. High-Intensity Interval Training (HIIT) has emerged as an effective strategy for reducing this detrimental FM. In 2016, AME2P laboratory was the first to demonstrate that HIIT training is more effective than continuous moderate-intensity training (MICT) in promoting the loss of intra-abdominal fat in postmenopausal women. A meta-analysis conducted by AME2P laboratory in 2018, including 39 scientific articles with 617 subjects, confirms the significant effects of HIIT on total and intra-abdominal fat loss in overweight or obese individuals . In addition to the tested modality (HIIT vs. MICT), it seems that the mode of locomotion (HIIT running vs. cycling) may impact body composition differently, with running being more effective for intra-abdominal fat loss and cycling for total FM loss. Cycling primarily involves concentric effort of the lower limbs, while running engages the lower limbs, trunk, and to a lesser extent, the upper limbs, involving both concentric and eccentric muscle contractions. These physiological/biomechanical differences have an impact on metabolic adaptations to exercise and recovery. Thus, at the same relative intensity during continuous exercise, oxygen consumption and energy expenditure are higher in running compared to cycling. Following exercises of intensity greater than 50% of VO2max, excess post-exercise oxygen consumption (EPOC) and lipid oxidation are higher in running compared to cycling. The greater muscle involvement (engaged muscle mass) and the eccentric nature of running (causing muscle damage) are likely responsible for these adaptations.

To better understand changes in body composition following HIIT training in running versus cycling among overweight or obese patients, the investigators propose to compare two isoenergetic HIIT sessions. The objective is to compare post-exercise (+2h) oxygen consumption and substrate utilization. Considering the influence of practice modalities on dietary compensations, the investigators will simultaneously measure spontaneous dietary intakes over the following 24 hours.

Objectives

The main objective is to compare two isoenergetic HIIT sessions: running vs. cycling.

The two tested modalities are as follows:

1. HIIT RUN: 9-12 x [45 seconds at 80% of HRmax followed by 1 minute 30 seconds of active recovery at a treadmill speed equivalent to 40% of HRmax].
2. HIIT BIKE: 9-12 x [45 seconds at 80% of HRmax followed by 1 minute 30 seconds of active recovery at a power equivalent to 40% of HRmax].

The theoretical maximum heart rate (HRmax) is calculated according to the formula of Gellish et al. (2007): HRmax = 207 - 0.7 x age.

The sessions are conducted in a random order. The second session is adapted (9-12 repetitions) to obtain isoenergetic exercises.

Through these modalities, the investigators will compare post-exercise oxygen consumption (during 2 hours) and carbohydrate and lipid oxidation during the exercise, the recovery period (during 2 hours) (MetaMax 3B Cortex, France), and the appetite 24hours post-exercise (from questionaniers and interview).

*Note that medical supervision of all participants is provided by the Health Department of the CREPS Auvergne-Rhône-Alpes in Vichy, which is authorized for such care. Physicians and physical activity professors are present on site.

General Hypotheses

The investigators propose the following hypotheses:

* Post-exercise oxygen consumption (2 hours) will be higher in HIIT running compared to cycling
* Higher post-exercise oxygen consumption following HIIT running could lead to an increase of lipid utilization during the recovery period.
* Energy intake over 24 hours will not differ due to the isoenergetic nature of the sessions.

ELIGIBILITY:
Inclusion Criteria:

- men with overweight or obesity (BMI between 25 kg/m2 and 35 kg/m2)

Exclusion Criteria:

* medical contraindications to intense physical activity,
* painful joints,
* taking ß-blocker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
oxygen consumption during the recovery period | Two hours after the end of the exercise
  Determination of oxygen consumption 2 hours after the exercise session (cycling and running). Determination from Metamax (3D Cortex).

SECONDARY OUTCOMES:
Lipid and carbohydrate oxidation during and after the exercise session (cycling and running). | Measurement during exercise and two hours after the end of the exercise
  Determination of lipid and carbohydrate oxidation during and after the exercise (HIIT cycling and running). Lipid and carbohydrate oxidation are measured from oxygen and carbon dioxide consumption (Metamax 3D Cortex).
Energy intakes 24 hours after the exercise | 24 hours post exercise
  evaluation of energy intakes after the exercise session (cycling vs running) during 24 hours (from questionnaires and interview)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Morel, Dr, Principal Investigator — CREPS Auvergne Rhône-Alpes / Vichy
Locations (1):
- CREPS Auvergne Rhône-Alpes / Vichy, Bellerive-sur-Allier, Allier, France